CLINICAL TRIAL: NCT00559507
Title: A Phase II Study of AZD0530 in Hormone Receptor-Negative, Metastatic or Unresectable, Locally Advanced Breast Cancer
Brief Title: Saracatinib in Treating Patients With Metastatic or Locally Advanced Breast Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00191; MSKCC-07112; N01CM62204 (NIH); N01CM62206 (NIH); CDR0000574281 (Registry Identifier: PDQ (Physician Database Query)); NCT01645605 (obsolete NCT alias); NCT01664481 (obsolete NCT alias)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2013-12

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Male Breast Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — saracatinib

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive saracatinib PO on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: saracatinib
  Other Names: AZD0530
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying saracatinib to see how well it works in treating patients with metastatic or locally advanced breast cancer that cannot be removed by surgery. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the disease control rate of AZD0530 (saracatinib) in patients with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To estimate the efficacy of AZD0530 in terms of overall response rate (complete and partial response) and progression free survival.

II. To describe the toxicity profile of AZD0530 in this patient population. III. To prospectively explore changes in circulating tumor cells from pre-treatment levels in patients receiving AZD0530.

OUTLINE:

Patients receive saracatinib orally (PO) on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the breast

  * Unresectable disease
  * Locally advanced or metastatic (American Joint Committee on Cancer [AJCC] stage IV) disease
* Estrogen receptor-negative and progesterone receptor-negative breast cancer defined as < 10% expression by immunohistochemistry (IHC)
* Measurable disease, defined (per Response Evaluation Criteria in Solid Tumors [RECIST]) as ≥ 1 unidimensionally measurable lesion ≥ 20mm by conventional techniques or ≥ 10 mm by spiral computed tomography (CT) scan

  * Measurable target lesions must not be in a previously irradiated field
* Patients with locally advanced, unresectable disease must have progression of disease following no more than one first-line chemotherapy regimen
* Patients with evidence of recurrent disease during or within 6 months after adjuvant chemotherapy will be considered to have failed one line of chemotherapy for metastatic disease
* Human epidermal growth factor receptor 2 (HER2)-positive patients, defined as immunohistochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) amplification > 2.1, must have received trastuzumab (Herceptin®) in either the adjuvant or metastatic setting and have had recurrence or progression of disease, respectively
* No known brain metastases
* Male and female patients eligible
* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2 (Karnofsky PS 60-100%)
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Urine protein creatinine (UPC) ratio must be ≤ 1.0

  * Patients with a UPC ratio > 1.0 must have a 24-hour urine protein < 1,000 mg to be eligible for study
* Not pregnant or nursing
* Women of child-bearing potential and men must use adequate contraception (e.g., hormonal or barrier method of birth control or abstinence) prior to, during, and for 8 weeks after completion of study therapy
* Able to understand and willing to sign a written informed consent document
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* No QTc interval ≥ 500 msecs
* No condition that impairs the ability to swallow AZD0530 tablets, including the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No intercurrent cardiac dysfunction including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
  * History of myocardial infarction within 6 months of treatment
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* No severe restrictive or obstructive lung disease according to baseline pulmonary function studies including any of the following pulmonary function test (PFT) parameters:

  * Total lung capacity < 60%
  * Forced vital capacity < 50%
  * Forced expiratory volume in one second (FEV_1) < 50%
  * Diffusion capacity of carbon monoxide (DLCO) < 50%
  * Resting room air O_2 saturation < 92% or a decline in O_2 saturation > 4% with exercise
* Patients with metastatic disease may have received no more than 1 prior chemotherapy regimen
* No unresolved toxicity ≥ grade 3 from agents received more than 3 weeks earlier
* No chemotherapy, radiotherapy, or investigational therapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study
* No luteinizing hormone-releasing hormone agonists within 4 weeks prior to study entry
* More than 7 days since prior and no concurrent use of specifically prohibited cytochrome P 450 3A4 (CYP3A4) agents
* No concurrent megestrol acetate, even when prescribed for appetite stimulation
* No other concurrent investigational or commercial agents for the treatment of breast cancer
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No concurrent megestrol acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Hudis, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 10/25/2007 Primary Compeltion Date 02/22/2011 Recruitment Location is medical clinic
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive saracatinib 175 mg PO on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 12
Completed | 9
Not Completed | 3
Not completed — Not treated, patient ineligible | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Saracatinib): Patients will receive AZD0530 175mg orally daily for 4 weeks.
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (38.18376618)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: DCR defined as complete response (CR), partial response (PR), stable disease (SD) > 24 weeks. Simon's two-stage optimal design was used to estimate the DCR of AZD0530 after 24 weeks of therapy since this design allowed for early termination of the study. Response and progression was evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions: Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: After 24 weeks of study therapy
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
participants | 0

2. Secondary Outcome: Overall Response Rate (CR and PR)
Description: Overall Response rate is defined as the sum of the complete response rate and partial response rate. Response and progression was evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions: Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: From start of treatment to 24 weeks after completion of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
participants
  Stable Disease | 3
  Progression of Disease | 6

3. Secondary Outcome: Median Time to Treatment Failure
Time Frame: From the start of treatment up to 4 weeks after completion of study treatment
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 9
Days | 82 [12 to 109]

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=9)
Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Adrenal insufficiency (General disorders) | 1 (1)
Sodium, low (hyponatremia) (General disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=9)
AST, SGOT (Blood and lymphatic system disorders) | 2 (2)
Fatigue (Metabolism and nutrition disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Glucose, high (hyperglycemia) (General disorders) | 1 (1)
Potassium, low (hypokalemia) (General disorders) | 1 (1)
Phosphate, low (hypophosphatemia) (General disorders) | 2 (2)
Bilirubin (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less